CLINICAL TRIAL: NCT04465084
Title: Assessment of Language Disorders in Multiple Sclerosis Patients
Acronym: LANSEP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Collaborators: Groupe Hospitalier Pitie-Salpetriere (Other); Saint Antoine University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: AGN_2020-18
Record Dates: First submitted 2020-07-02; First posted 2020-07-09 (Actual); Last update posted 2023-02-15 (Actual); Status verified 2023-02

CONDITIONS: Sclerosis; Language Disorders
MeSH Terms: conditions — Sclerosis; Language Disorders

STUDY DESIGN:
Intervention Model Description: Relapsing-Remitting Multiple Sclerosis and Secondary Progressive Multiple Sclerosis.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Case (Other): Relapsing-Remitting Multiple Sclerosis and Secondary Progressive Multiple Sclerosis.
  Interventions: Other: Case
- Witness (Other): Person matched to a "case" on age (+/-3 years) and education level
  Interventions: Other: Withness

INTERVENTIONS:
Other: Case — Battery of standardised and normalised tests evaluating different cognitive functions Experimental language tasks MRI
  Arms: Case
Other: Withness — Experimental language tasks MRI
  Arms: Witness

SUMMARY:
Multiple sclerosis (MS) is an autoimmune disease of the central nervous systems that results in focal inflammatory lesions and then diffuse and degenerative inflammatory phenomena. It is considered to be the leading cause of non-traumatic disability in young adults.

Cognitive impairment is a common and disabling part of MS. Studies carried out in the years 1990-2000 estimated their frequency to be between 40 and 60% of MS patients: they reflect the natural history of the disease. Effective treatments for the inflammatory component of the disease that are now available may have led to a reduction in their frequency.

Cognitive disorders were identified at an early stage of the disease and affect certain areas preferentially:

* The most common achievement is the reduction in the speed of information processing. It is present from the early stage of the disease. Progressive deterioration over time is observed, which is a prognostic factor for long-term cognitive decline.

Long-term memory was impaired in 40-65% of patients in historical cohorts. More specifically, encoding and retrieval were affected, with storage and consolidation being preserved.

* The attainment of executive functions is also common.
* Phonemic and semantic fluency are also disturbed in MS patients. Among cognitive impairments, language impairment has been little studied in MS: in 2016 only 22 controlled studies were identified. The assessments carried out were most often partial, making it impossible to define the characteristics or to conclude that specific linguistic impairments are independent of other cognitive impairments. Finally, recent studies suggest that the frequency of language impairment in MS may be underestimated.

Therefore, it seems important to assess the prevalence of language disorders in a large cohort of patients with RRMS or MS, and to characterize these disorders by identifying the linguistic processes involved and the brain substrates involved. This will make it possible to envisage the implementation of more systematic screening for language disorders in MS and to improve patient management, in particular by developing targeted rehabilitation protocols.

DETAILED DESCRIPTION:
Relapsing-Remitting Multiple Sclerosis and Secondary Progressive Multiple Sclerosis.

Experimental tasks based on psycholinguistics and functional MRI are not standardized tests. To be able to interpret the results of patients, they must therefore be compared with healthy controls of the same age (+/-3 years) and level of education.

This study will require the inclusion of cases and controls matched to these cases on the above characteristics.

Patients who are seen in consultation or day hospitalization and who meet the inclusion and non-inclusion criteria will be offered the opportunity to participate in the study. Accompanying persons accompanying patients "matching" with included patients who meet the inclusion and non-inclusion criteria will also be offered the opportunity to participate in the study.

Inclusion visit (D0) :

* Completion of the HAD self-questionnaire
* Validation of inclusion and exclusion criteria
* Signature of consent
* Collection of socio-demographic data to adjust standardized test results (age, gender, socio-economic and education level)
* Completion of the computerized ECVB self-questionnaire with the help of a clinical research technician: only for cases
* Scheduling of the HDJ assessment day (maximum 6 months after the inclusion visit)

Visit 1 (assessment in HDJ) (D0 + 6 months maximum) :

* Neurological examination of the patient and performance of an EDSS if necessary
* Battery of standardised and normalised tests evaluating different cognitive functions (Annexes 1 and 2 to 9): only for cases
* Experimental language tasks (see description in section 6): for cases and controls
* Non-injected structural and functional encephalic MRI: only for cases with language impairment detected in the examination battery (and their matched controls)

ELIGIBILITY:
Criteria for inclusion of cases :

* Patient with a diagnosis of RRMS or MS according to the Mac Donald criteria 2017
* Patient between 18 and 60 years old inclusive
* Express consent to participate in the study
* Affiliate or beneficiary of a social security scheme
* Patients in structured computerised databases for MS

Criteria for non-inclusion of cases

* Pregnant or breastfeeding woman
* Patient with a psychological disorder that may induce a language disorder (AHH - anxiety score ≥ 8 or AHH - depression score ≥ 8) (scale in Appendix 11)
* Patient with a history of language impairment before the onset of MS
* Patient receiving speech therapy for language disorders
* Patient whose mother tongue is not French
* Patient with too much dysarthria hindering the intelligibilité́ of his words
* Patient with uncorrected visual and/or hearing impairment
* Neurological diseases (other than MS)
* Psychiatric disorders
* Contraindication to MRI (claustrophobia, implanted equipment such as pacemaker).

Criteria for inclusion of witnesses

* Person matched to a "case" on age (+/-3 years) and education level (see Annex 11)
* Express consent to participate in the study
* Affiliate or beneficiary of a social security scheme

Criteria for non-inclusion of witnesses

* Pregnant or breastfeeding woman
* Psychic disorder that can induce a language disorder (AHH - anxiety score ≥ 8 or AHH - depression score ≥ 8) (Appendix 10)
* History of Language Impairment
* Person receiving speech therapy for language disorders
* Person whose mother tongue is not French
* Person with too much dysarthria hindering the intelligibilité́ of his words
* Uncorrected visual and/or hearing impairment
* Person with a neurological disease
* Psychiatric disorders
* Contraindication to MRI (claustrophobia, implanted equipment such as pacemaker).

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 142 (Actual)
Dates: Start 2020-08-17 (Actual); Primary Completion 2020-08-17 (Actual); Study Completion 2022-07-08 (Actual)

PRIMARY OUTCOMES:
proportion de patient with language disorders in patients with RRMS or MS | 6 month

CONTACTS AND LOCATIONS:
Locations (1):
- Antoine GUEGUEN, Paris, France

IPD SHARING:
Plan to Share IPD: No